CLINICAL TRIAL: NCT06550947
Title: Immunohistochemical Expression and Prognostic Significance of ALDOA in Bladder Urothelial Carcinoma.
Brief Title: ALDOA Expression in Bladder Urothelial Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Hesham John, Demonstrator, Assiut University
Other Study IDs: Bladder immunohistochemistry
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bladder Urothelial Carcinoma
MeSH Terms: interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Immunohistochemistry — Immunohistochemical expression of ALDOA in bladder urothelial carcinoma

SUMMARY:
1. Study the immunohistochemical expression of ALDOA in bladder urothelial cancer.
2. Correlate between ALDOA expression in specimens and different cilnicopathological factors.
3. Correlate between ALDOA expression and urothelial cancer prognosis and survival.

DETAILED DESCRIPTION:
Bladder cancer is the 7th most prevalent malignancy and the 13th cause of cancer related death worldwide1. In Egypt, it's the third most common tumor2.

The most common histologic subtype of bladder cancer is urothelial carcinoma3. Bladder cancer is divided according to absence or presence of muscle invasion into non-muscle invasive bladder cancer and muscle invasive bladder cancer 3.

Despite the advance in diagnosis and development of therapeutic options of urothelial cancer, the recurrence and progression rate remains high4.

The conventional histopathological evaluation of urothelial cancer is vital for diagnosis and prediction of patient's prognosis. However, it doesn't fully reflect the biological behavior of the tumor or the clinical outcome of the patient5.

Under hypoxic conditions, cancer cells produce ATP by glycolysis, which provide energy for tumor proliferation and dissemination6,7. Glycolytic enzymes are abnormally activated in cancer cells8,9. Thus, several studies have identified glycolytic enzymes or related metabolic pathways as potential drug targets. One of the typical glycolytic enzymes is Aldolase A (ALDOA) 6 which is the most abundant glycolytic enzyme detected in tumors10.

Several studies have identified ALDOA as an oncogene in different types of malignancy 6,8,10-12. The oncogenic potential of ALDOA contributed to its ability to stimulate DNA synthesis and accelerate S phase in tumor cell cycle6-8.

In addition, studies have shown that ALDOA promotes tumor cell invasion by negative regulation of E-cadherin and by activation of MAPK, AKT and EGFR signaling pathways7,11,13.

Thus, increased expression of ALDOA in tumor predicts a bad prognosis and poor survival of patients13-15.

ELIGIBILITY:
Inclusion Criteria:

* All cases diagnosed as bladder urothelial cancer with known follow-up data and presence of muscle proper detected in the specimens.

Exclusion Criteria:

1. Subtypes of bladder cancer other than urothelial carcinoma subtype.
2. Cases of urothelial carcinoma without known follow up data.
3. Cases of urothelial carcinoma without muscle proper detected in the specimen.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted using formalin fixed paraffin embedded blocks of fifty cases of urothelial carcinomas . These blocks will be obtained from laboratory archives of the Pathology Department, Assiut University Hospital, Faculty of Medicine. Clinical data for this study will be obtained from laboratory archives of the pathology department, Assiut University Hospital, Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the immunohistochemical expression of ALDOA in bladder urothelial carcinoma. | Baseline
  Microscopic examination of bladder urothelial carcinoma spicemens and staining them with ALDOA marker

SECONDARY OUTCOMES:
Evaluate relation between ALDOA expression and cilnicopathological features and patient survival. | Baseline
  Correlate between ALDOA expression and the different clinicopathological factors of patients and their survival.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Elsers, Professor, Study Director — Head of Pathology Department

REFERENCES:
- See also: Related Info — https://mjcu.journals.ekb.eg/article_295963.html
- See also: Related Info — https://www.menoufia-med-j.com/journal/vol31/iss3/17/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10272547/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9720515/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC11260772/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5993145/
- See also: Related Info — https://www.annualreviews.org/content/journals/10.1146/annurev-cancerbio-030518-055425
- See also: Related Info — https://www.nature.com/articles/s41419-019-1968-4
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10344634/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9556458/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31081974/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5338975/
- See also: Related Info — https://www.nature.com/articles/s41598-022-15866-4